CLINICAL TRIAL: NCT01420432
Title: Phase II Study of Umbilical Cord/Placenta-Derived Mesenchymal Stem Cells to Treat AS
Brief Title: Safety and Efficacy Study of Umbilical Cord/Placenta-Derived Mesenchymal Stem Cells to Treat Ankylosing Spondylitis (AS)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Chengyun Zheng, Department of Hematology of the 2nd Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zhangni
Record Dates: First submitted 2011-08-11; First posted 2011-08-19 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-04

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Umbilical Cord/placenta-Derived MSC; Transplantation
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human umbilical cord-derived MSCs and DMARDs (Experimental): Human umbilical cord-derived MSCs at a dose of 1.0E+6 MSC/kg, repeated after three months and DMARDs such as sulfasalazine,methotrexate,thalidomide po for 12 months
  Interventions: Biological: Human umbilical cord-derived MSCs
- DMARDs (No Intervention): DMARDs such as sulfasalazine,methotrexate,thalidomide po for 12 months

INTERVENTIONS:
Biological: Human umbilical cord-derived MSCs — 1.0E+6 MSC/kg, IV drop and repeat repeated after three months
  Arms: Human umbilical cord-derived MSCs and DMARDs

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mesenchymal stem cells (MSCs) derived from human umbilical cord/placenta at a dose of 1.0E+6 MSC/kg in subject for the therapy of Ankylosing spondylitis (AS)

DETAILED DESCRIPTION:
Ankylosing spondylitis (AS) is a chronic, progressive inflammatory rheumatic disease involving primarily the sacroiliac joints and the axial skeleton. The main clinical features are back pain and progressive stiffness of the spine. Oligoarthritis of the hips and shoulders, enthesopathy, and anterior uveitis are common, and involvement of the heart and lungs is rare. The current understanding of the pathogenesis of this disorder is limited.It mainly about to hereditary susceptibility (eg hla-b27),infection and autoimmunity.

Although traditional drugs, such as Nonsteroidal antiinflammatory drugs (NSAIDs) disease-modifying antirheumatic drugs (DMARDs such as MTX,SASP OR thalidomide) and steroids have been used in the treatment of AS, however, many studies have indicated that the overall response to these drugs is not satisfied. Addition, the severe side effects of these drugs have also been observed. The management of AS patients therefore remains unsatisfactory and targeted therapies are needed. Human MSCs isolated from human umbilical cord/placenta have been shown to have immunoregulatory, immunosuppressive, stimulating hematopoiesis and tissue repairing properties. This study will evaluate the safety and effectiveness of MSC transplantation in the AS patients.

This study will last 2 to 3 years. Participants will be randomly assigned to receive either MSC transplant +DMARDs therapy (experimental group) or DMARDs therapy (control group). Patients will undergo MSC transplant at the start of the study on Day 0. After 3 months, patients will receive the second MSC transplantation. After six and twelve months from the first transplantation, patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 18~60 years old with plan to infuse MSCs.
2. Diagnosis of "Definite AS" (arthritis of the spine) as defined by the modified New York criteria
3. Stable doses of sulfasalazine,methotrexate,thalidomide,hydroxychloroquine, low-dose corticosteroids, and NSAIDs are permitted
4. Patients must have an ECOG 0~2.
5. No moderate or sever organ dysfunction: Ejection fraction>45%; Creatinine <176 umol/L.
6. No severe infection.
7. Each patient must sign written informed consent.

Exclusion Criteria:

1. Other serious concomitant diseases (uncontrolled/severe kidney, liver, haematological, gastrointestinal, endocrine, cardiovascular, pulmonary, neurological or cerebral disease)
2. Psychiatric condition that would limit informed consent.
3. HIV, hepatitis B or C, tuberculosis, other infections
4. Positive Pregnancy Test or lactation
5. Patient has enrolled another clinical trial study within last 4 weeks.
6. Contraindications to MSC

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The Assessment of Spondyloarthritis International Society (ASAS)20 response | 1 year
  ASAS measures symptomatic improvement in AS patients.ASAS=4 domains:patient global assessment of disease activity,pain,function,inflammation.ASAS 20=20% improvement(vs.baseline)and an abosolute change≥1 units on a 0-10 scale(0=no disease activity;10=high disease activity)for ≥3 domains,and no worsening in remaining domain.
  Patient global Pain Function (as measured by the Bath Ankylosing Spondylitis Functional Index - BASFI) Inflammation (mean of the Bath Ankylosing Spondylitis Disease Activity Index - BASDAI question 5 and 6)
erythrocyte sedimentation rate (ESR) | 1 year
  erythrocyte sedimentation rate (ESR) level will be mainly observed after transplanting 3, 6,12-month.
imageology | 1 year
  imageology will be mainly observed after transplanting 3, 6,12-month.
C-reactive protein (CRP) | 1 year
  C-reactive protein (CRP) level will be mainly observed after transplanting 3, 6,12-month.

SECONDARY OUTCOMES:
Percentage of systemic T regulatory cell population | 1 year
  Percentages of T regulatory cell population in peripheral blood will be tested in every 3 months after transplanting MSCs for one year
Side effects | 1 year
  Side effects were observed after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: chengyun zheng, Ph. D, Principal Investigator — Department of Hematology of The 2nd Hospital of Shandong University
Locations (1):
- Department of Hematology of the 2nd Hospital of Shandong University, Jinan, Shandong, China